CLINICAL TRIAL: NCT06671262
Title: Neoadjuvant Toripalimab and Radiotherapy Treatment in Lymph Nodes Positive HR Positve Breast Cancer（NEOTRIO-HR）
Brief Title: Neoadjuvant Toripalimab and Radiotherapy Treatment in N+ HR+ Breast Cancer
Acronym: NEOTRIO-HR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y2024-0857
Record Dates: First submitted 2024-10-10; First posted 2024-11-04 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Breast Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The control group (Active Comparator): Patients in this arm receive only a single injection of toripalimab without any radiotherapy as an initial treatment. After a three-week interval, patients receive the standard neoadjuvant chemotherapy in combination with toripalimab, starting with four cycles of paclitaxel and toripalimab, followed by four cycles of epirubicin and toripalimab.
  Interventions: Drug: Immuno-chemotherapy
- The SBRT-combined group 1 (Experimental): Patients enrolled in this treatment arm will undergo SBRT focused on the primary tumor, receiving a total dose of 24Gy divided into three fractions over the course of 3 to 5 working days. Following the radiation therapy, toripalimab will be administered between the second and fifth days post-treatment. After a three-week rest period, patients will commence the standard neoadjuvant chemotherapy regimen combined with toripalimab. This regimen will begin with four cycles of paclitaxel combined with toripalimab and followed by four cycles of epirubicin combined with toripalimab.
  Interventions: Radiation: SBRT; Drug: Immuno-chemotherapy
- The SBRT-combined group 2 (Experimental): In this treatment protocol, patients will receive a total radiation dose of 24Gy in three fractions, specifically targeting the primary tumor. Concurrently, the axillary lymph nodes will be treated with a dose of 9Gy in three fractions. This radiation therapy will be conducted over a period of 3 to 5 working days. Following the radiation therapy, toripalimab will be administered between the second and fifth days after the completion of the radiation treatment. After a three-week interval, patients will proceed with the standard neoadjuvant chemotherapy regimen combined with toripalimab. This regimen includes an initial phase of four cycles of paclitaxel paired with toripalimab, which will be followed by a subsequent phase of four cycles of epirubicin paired with toripalimab.
  Interventions: Radiation: SBRT; Drug: Immuno-chemotherapy

INTERVENTIONS:
Radiation: SBRT — Target the primary tumor region with a single dose of 8Gy, or deliver a dose of 3Gy to the axillary lymph nodes, administered once a day for three consecutive days.
  Arms: The SBRT-combined group 1; The SBRT-combined group 2
Drug: Immuno-chemotherapy — Standard new adjuvant treatment with toripalimab combined with chemotherapy, that is in the first phase consisting of paclitaxel and toripalimab for four cycles, followed by epirubicin, cyclophosphamide, and toripalimab for another four cycles.

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety in patients with lymph node-positive HR+/HER2- breast cancer. The main questions it aims to answer are:

* Can the incorporation of intensified radiation to the tumor (tumor boost) enhance the pCR rate on the basis of neoadjuvant immuno-chemotherapy？
* Can it improve the level of residual cancer burden (RCB) and change the tumor immune microenvironment? and How safe will be the combined therapy?

Participants will be randomly assigned to one of three treatment regimens:

1. Preoperative toripalimab combined with SBRT targeting both the primary tumor and axillary lymph nodes, followed by chemotherapy;
2. Preoperative toripalimab combined with SBRT focused solely on the primary tumor, followed by chemotherapy;
3. Preoperative toripalimab combined with chemotherapy alone.

Following the completion of their respective treatment regimens, participants will proceed to undergo surgery. The effectiveness of the treatments will be assessed through pathological evaluations, as well as by measuring levels of residual cancer burden (RCB) and examining changes in the tumor immune microenvironment.

The study aims to evaluate the safety of these combined treatment approaches and to determine if they offer superior efficacy compared to outcomes reported in previous studies.

DETAILED DESCRIPTION:
Breast cancer is a leading malignancy among women globally, with early diagnosis and treatment being crucial for better outcomes. Over 90% of breast cancer patients are diagnosed at an early stage, and approximately two-thirds have the hormone receptor-positive/human epidermal growth factor receptor 2-negative (HR+/HER2-) subtype. Despite this, these patients often exhibit resistance to neoadjuvant chemotherapy, with a pathologic complete response (pCR) rate of only 5-15%, which is significantly lower compared to other subtypes and is associated with poor prognosis. This indicates the necessity for optimizing current treatment strategies.

In recent years, significant advancements have been made in the application of immunotherapy for breast cancer. The studies demonstrated that the addition of immune checkpoint inhibitors to neoadjuvant chemotherapy for patients with high-risk early-stage HR+/HER2- breast cancer significantly improved pCR rates.

Building on these findings, this study proposes a novel strategy of dose-intensified radiation to the tumor (tumor boost) during the neoadjuvant immuno-chemotherapy phase. The advantage of this approach is that it can activate the immune system while the tumor tissue is still intact, providing a rich source of tumor antigens, which aids in enhancing the immune system's recognition and destruction of cancer cells.

Toripalimab is an optimal immunotherapy agent to study, as this agent has recently been approved by the FDA for use in multiple tumor types. It is therefore ready to be tested for efficacy in other disease sites and in combination with other treatments. This study will provide valuable insights into the potential of immunotherapy in combination with radiotherapy to improve outcomes for patients with lymph nodes-positive, high-risk HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* High-risk HR+/HER2-negative breast cancer is defined as ER≥1%, HER2-negative (<2+ Her2 IHC or <2.2 HER2/CEP17 ratio by FISH) and either histologic grade II-III or a high-risk genomic assay score (Oncotype RS>25, high risk Mammaprint, PAM-50, EndoPredict or ProSigna score). primary tumor size ≥1.0 cm in maximum diameter and axillary node-positive breast cancer;
* Stage T1-4N+M0 (i.e., Stage II, III), with confirmed N+ by biopsy, and no signs of distant metastasis;
* The initial PD-L1 expression level conducted on the tumor tissue sample with Combined Positive Score (CPS) or Tumor Proportion Score (TPS)< 10%;
* ECOG score of 0-1;
* Screening laboratory values must meet the following criteria: i. White blood cells (WBCs) ≥ 2000/μL ii. Absolute neutrophil count (ANC) ≥ 1500/μL iii. Platelets ≥ 100 x 103/μL iv. Hemoglobin ≥ 11.0 g/dL v. Serum creatinine ≤ 2 mg/dL (or glomerular filtration rate ≥ 40 ml/min) vi. AST ≤ 2.5 x upper limit of normal (ULN) vii. ALT ≤ 2.5 x ULN viii. Total bilirubin within normal limits (except subjects with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL) ix. INR ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulant(s) x. Negative HIV screening test xi. Negative screening tests for Hepatitis B and Hepatitis C. Patients with positive results that do not indicate true active or chronic infection may enroll after discussion and consensus agreement by the treating physician and principal investigator.

Exclusion Criteria:

* Inflammatory breast cancer
* Life-threatening organ dysfunction or complications, active infectious diseases, active hepatitis B, hepatitis C virus infection, autoimmune diseases within two years, undergoing immunosuppressive drug treatment or chronic systemic corticosteroid therapy (dose exceeding 10mg per day of prednisone or equivalent);
* Clinically symptomatic heart disease;
* Previous systemic treatment or radiotherapy for breast cancer;
* Patients with cosmetic breast implants, i.e., having implants under the skin at the time of diagnosis;
* Radiotherapy contraindications: history of radiotherapy;
* Women shall not be breastfeeding.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 74 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | At the end of immuno-chemotherapy up to 4-6 months
  Pathological Complete Response (pCR) is characterized by the absence of any invasive residual primary tumor in both the breast and lymph nodes. The primary objective of this study is to compare the pCR rates between two treatment approaches: neoadjuvant toripalimab combined with SBRT followed by immuno-chemotherapy, and neoadjuvant toripalimab combined with chemotherapy.

SECONDARY OUTCOMES:
RCB level | breast surgery up to 4-6 months after trial initiation
  Residual Cancer Burden (RCB) level is a classification system used to assess the amount of cancer remaining in the breast tissue and lymph nodes after neoadjuvant chemotherapy. It is determined by evaluating several factors including the primary tumor area, the percentage of the tumor area that is invasive cancer, and the extent of lymph node involvement. The RCB index categorizes patients into four groups from group 0 to III indicating none to extensive residual cancer burden.
TILs | Pre-treatment, post-initial dose of Toripalimab with or without radiation up to 4 weeks, and at surgical resection up to 4-6 months.
  Changes in the tumor-infiltrating lymphocyte score (TILs), as determined by the Salgado criteria, indicate an engagement of the immune system in cancer, with scores ranging from 0 to 100%. A higher score in TILs correlates with improved patient outcomes. The planned collection of biopsy samples at three critical points-before treatment, after the initial dose of Toripalimab with or without radiation therapy, and at the time of surgical resection-will enable a comprehensive serial evaluation of TILs. This approach will help to quantify the impact of radiation therapy on the immune response induced by Toripalimab.
SBRT-related Adverse Events | at least once a week within 2-4 weeks after the start of radiotherapy.
  Treatment toxicities. radiation-related AEs, especially Acute Radiation Dermatitis.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China